CLINICAL TRIAL: NCT00462540
Title: A Crossover Study in the Treatment of Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director, Clinical Affairs, Dey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201-081
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Formoterol; Ipratropium; Crossover
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium; Albuterol

INTERVENTIONS:
Drug: Formoterol Fumurate inhalation solution 20 mcg
Drug: Ipratropium bromide 18 mcg and albuterol sulfate 103 mcg

SUMMARY:
The purpose of this study is to compare the efficacy of Formoterol Fumarate Inhalation Solution (FFIS) 20 mcg BID to Combivent® Inhalation Aerosol [2 inhalations from metered dose inhaler (MDI)of 18 mcg ipratropium bromide and 103 mcg albuterol sulfate QID], and to Compare the preference/compliance of BID nebulization to QID use of MDI

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Smoker or exsmoker with at least 10 years smoking at least one pack of cigarettes per day
* Meet lung function requirements

Exclusion Criteria:

* Diagnosis of Asthma
* Significant disease other than COPD
* Female pregnant or lactating or planning to become pregnant

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Lung function after 2 weeks of treatment

SECONDARY OUTCOMES:
Lung function at each time point, patient questionnaires, medication compliance,
adverse events, clinical labs, vital signs, ECGs, physical exams

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Research Site, San Diego, California
  - Research Site, Denver, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Panama City, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Sunset, Louisiana
  - Research Site, Charlotte, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Gaffney, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Johnson City, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Spokane, Washington
  - Research Site, Morgantown, West Virginia

REFERENCES:
- [Result] Sutherland ER, Brazinsky S, Feldman G, McGinty J, Tomlinson L, Denis-Mize K. Nebulized formoterol effect on bronchodilation and satisfaction in COPD patients compared to QID ipratropium/albuterol MDI. Curr Med Res Opin. 2009 Mar;25(3):653-61. doi: 10.1185/03007990802708152. PMID 19232039